CLINICAL TRIAL: NCT03830437
Title: Salivary Cortisol as Stress Marker in Newborns Subjected to Double Weighing With Body Weight Loss of 3±1,5% at 24 hr From Birth
Brief Title: Salivary Cortisol as Stress Marker in Newborns Subjected to Double Weighing With Physiological Body Weight
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernando, Chief of NICU, Fondazione Poliambulanza Istituto Ospedaliero
Other Study IDs: 3175
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cortisol Overproduction
Keywords: Newborn; Salivary Cortisol Level; Double Weghing; Physiological weight loss; Breastfeeding; Stress marker
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: The group will be subjected to double weighing, before and after the next 6 breastfeeding. Breastfeeding will be carried out each 4 hr.
  Interventions: Other: Evaluation of newborn stress; Other: Evaluation of body weight trend
- Control group: The group will be subjected to monitoring of body weight only at 24, 36 hr and 48 hr of life.
  Interventions: Other: Evaluation of newborn stress; Other: Evaluation of body weight trend

INTERVENTIONS:
Other: Evaluation of newborn stress — Newborn stress will be evaluated by salivary cortisol levels at 48 hr of life. Saliva sample of the newborns will be collected in oral cavity at 48 hr of life. Samples collected will be storage at -80 C for up to 4 months and analysed by analysis laboratory of Poliambulanza Foundation.
Other: Evaluation of body weight trend — Body weight trend between newborns subjected to double weighing or to body weight control will be carried out at 36 hr and 48 hr of life

SUMMARY:
According to scientific revisions, salivary cortisol is a valid method for measuring adrenocortical activity in newborns because it is non-invasive in fact the measurement of salivary cortisol has been used as a stress marker in newborns since 1992. The mechanism by which cortisol induces stress, concerns the hypothalamic-pituitary-adrenal axis. The hypothalamus produces the corticotropin-releasing hormone, which stimulates the production of adrenocorticotropin by hypophysis. Adrenocorticotropin induces the secretion of glucocorticoids such as cortisol by stimulating the cortex of the adrenal gland. An appropriate release of cortisol due to stress factor is vital for surviving and the loss of this mechanism increase the risk of morbidity and mortality for newborns. However, prolonged exposure to a high level of cortisol may increase the risk of cognitive and behavioural disorders, hypertension, hyperlipidaemia, insulin resistance, immune deficiency and hippocampal impairment. The separation from the mother, the exposure to painful procedures but also routine interventions such as physical examination, diaper changes and bathing increase the salivary cortisol level of the newborn compared to the basal state. The measurement of salivary cortisol in the newborn therefore has the aim of understanding and preventing those stressful conditions that may have long-term side effects. For this reason, the lose weight in the first days and double weighing should be a stress practice for the newborn.

DETAILED DESCRIPTION:
After the phase of early adaptation, newborn must learn quickly to live out of the mother uterus. In this phase of life, physiological mechanisms are activated. Newborn loss body weight because loss liquid by respiration, feces, urine and not adequate feeding. Body weight loss after birth is physiological when is lower than 10% but is also important the evaluation of body weight daily trend that must be lower than 5%. If newborn shows physiological body weight loss, no treatment will be necessary and rooming-in can continue together with exclusively breastfeeding.

Furthermore, if newborn lose more than 10% of body weight during 48hr of life or more than 5% of body weight in a day, a dehydration state will occur that will influence negatively the physiological cardio-circulatory and kidney adaptation. In these cases, is important execute controls and a specific therapy. When body weight loss is between 7%-10%, usually in Neonatology wards it is used double weighing before and after breastfeeding. This practice evaluates colostrum quantity that is assumed from infant during feeding and the necessity of milk formula integration to prevent an excessive body weight loss. Diuresis is also monitored, and parents are informed on the benefits of breastfeeding.

If body weight loss is greater than 10%, diuresis is monitored weighing the diaper and haematological examinations are performed. In this case, it is counselled an artificial milk integration after breastfeeding. Discharge can be influenced from the results of the controls and must be executed for the security of the newborn.

Health care providers must not be underestimated the possible allergies to formula milk and the mothers that give up breastfeeding after the use of formula milk. The newborn should receive breastfeeding from the delivery room. It is good practice, when the milk secretion is enough, to attach the infant to a single breast for each feeding and let it suck for 15-20 minutes. Quantity of milk that newborn assume for each feeding is object of careful evaluation. Double weighing consists in weighing newborn before and after feeding: the body weight difference is the quantity of milk assumed. In the first day of life, newborn should suck 10 gr of colostrum or milk for each feeding. Then starting from the second day of life, the quantity of milk assumed must be increased of 10 gr/die for the first week.

According to scientific revisions, salivary cortisol is a valid method for measuring adrenocortical activity in newborns because it is non-invasive in fact the measurement of salivary cortisol has been used as a stress marker in newborns since 1992. The mechanism by which cortisol induces stress, concerns the hypothalamic-pituitary-adrenal axis. The hypothalamus produces the corticotropin-releasing hormone, which stimulates the production of adrenocorticotropin by hypophysis. Adrenocorticotropin induces the secretion of glucocorticoids such as cortisol by stimulating the cortex of the adrenal gland. An appropriate release of cortisol due to stress factor is vital for surviving and the loss of this mechanism increase the risk of morbidity and mortality for newborns. However, prolonged exposure to a high level of cortisol may increase the risk of cognitive and behavioural disorders, hypertension, hyperlipidaemia, insulin resistance, immune deficiency and hippocampal impairment. The separation from the mother, the exposure to painful procedures but also routine interventions such as physical examination, diaper changes and bathing increase the salivary cortisol level of the newborn compared to the basal state. The measurement of salivary cortisol in the newborn therefore has the aim of understanding and preventing those stressful conditions that may have long-term side effects. For this reason, the lose weight in the first days and double weighing should be a stress practice for the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 37-42 wks
* Body Weight: >2500 g
* Body weight loss >3±1,5% at 24 hr from birth
* First-born
* Eutocic delivery
* Mother BMI:19-24
* Glycaemia >50 mg/dl

Exclusion Criteria:

* Mother disease
* Admission in NICU
* Neonatal pathologies
* Utilization of human milk
* Body weight loss > 10%

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Caucasian newborns with 37-42 weeks of gestational age and that live in Lombardia.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of salivary cortisol levels | 48 hours
  Evaluation of salivary cortisol level as stress marker in newborns with body weight loss of 3±1,5% at 24 hours from birth subjected to double weighing or to body weight control at 36 hours and 48 hours of life.

SECONDARY OUTCOMES:
Evaluation of body weight trend | 48 hours
  Evaluation of body weight trend between newborns subjected to double weighing or to body weight control at 36 hours and 48 hours of life.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, M.D., Principal Investigator — Fondazione Poliambulanza Istituto Ospedaliero; Laura Linetti, Dott., Study Director — Fondazione Poliambulanza Istituto Ospedaliero
Locations (1):
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janet M. Rennie, "Textbook of Neonatology" Elsevier Health Sciences, London, 2012
- [Background] Horta, B.L.; Victora, C.G. Long-Term Effects of Breastfeeding: A Systematic Review; World Health Organization: Geneva, Switzerland, 2013, pp. 1-68
- [Result] Rodriguez G, Ventura P, Samper MP, Moreno L, Sarria A, Perez-Gonzalez JM. Changes in body composition during the initial hours of life in breast-fed healthy term newborns. Biol Neonate. 2000;77(1):12-6. doi: 10.1159/000014189. PMID 10658825
- [Result] Thulier D. Weighing the Facts: A Systematic Review of Expected Patterns of Weight Loss in Full-Term, Breastfed Infants. J Hum Lact. 2016 Feb;32(1):28-34. doi: 10.1177/0890334415597681. Epub 2015 Aug 7. PMID 26253288
- [Result] Noel-Weiss J, Courant G, Woodend AK. Physiological weight loss in the breastfed neonate: a systematic review. Open Med. 2008;2(4):e99-e110. Epub 2008 Oct 28. PMID 21602959
- [Result] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Result] Flaherman VJ, Kuzniewicz MW, Li S, Walsh E, McCulloch CE, Newman TB. First-day weight loss predicts eventual weight nadir for breastfeeding newborns. Arch Dis Child Fetal Neonatal Ed. 2013 Nov;98(6):F488-92. doi: 10.1136/archdischild-2012-303076. Epub 2013 Jul 17. PMID 23864443
- [Result] Bertini G, Breschi R, Dani C. Physiological weight loss chart helps to identify high-risk infants who need breastfeeding support. Acta Paediatr. 2015 Oct;104(10):1024-7. doi: 10.1111/apa.12820. Epub 2014 Oct 22. PMID 25283590
- [Result] Ferrandez-Gonzalez M, Bosch-Gimenez V, Lopez-Lozano J, Moreno-Lopez N, Palazon-Bru A, Cortes-Castell E. Weight loss thresholds to detect early hypernatremia in newborns. J Pediatr (Rio J). 2019 Nov-Dec;95(6):689-695. doi: 10.1016/j.jped.2018.06.005. Epub 2018 Jul 18. PMID 30030986
- [Result] Righard L, Alade MO. Effect of delivery room routines on success of first breast-feed. Lancet. 1990 Nov 3;336(8723):1105-7. doi: 10.1016/0140-6736(90)92579-7. PMID 1977988
- [Result] Jang GJ, Kim SH, Jeong KS. [Effect of postpartum breast-feeding support by nurse on the breast-feeding prevalence]. Taehan Kanho Hakhoe Chi. 2008 Feb;38(1):172-9. doi: 10.4040/jkan.2008.38.1.172. Korean. PMID 18323730
- [Result] Woolridge MW, Baum JD, Drewett RF. Individual patterns of milk intake during breast-feeding. Early Hum Dev. 1982 Dec 6;7(3):265-72. doi: 10.1016/0378-3782(82)90089-5. PMID 7160336
- [Result] Cignacco E, Denhaerynck K, Nelle M, Buhrer C, Engberg S. Variability in pain response to a non-pharmacological intervention across repeated routine pain exposure in preterm infants: a feasibility study. Acta Paediatr. 2009 May;98(5):842-6. doi: 10.1111/j.1651-2227.2008.01203.x. Epub 2009 Jan 13. PMID 19183121
- [Result] De Bernardo G, Riccitelli M, Giordano M, Proietti F, Sordino D, Longini M, Buonocore G, Perrone S. Rooming-in Reduces Salivary Cortisol Level of Newborn. Mediators Inflamm. 2018 Mar 8;2018:2845352. doi: 10.1155/2018/2845352. eCollection 2018. PMID 29706798
- [Result] Levine S. Developmental determinants of sensitivity and resistance to stress. Psychoneuroendocrinology. 2005 Nov;30(10):939-46. doi: 10.1016/j.psyneuen.2005.03.013. PMID 15958281
- [Result] Morelius E, Theodorsson E, Nelson N. Salivary cortisol and mood and pain profiles during skin-to-skin care for an unselected group of mothers and infants in neonatal intensive care. Pediatrics. 2005 Nov;116(5):1105-13. doi: 10.1542/peds.2004-2440. PMID 16263996
- [Result] Gunnar MR, Talge NM, Herrera A. Stressor paradigms in developmental studies: what does and does not work to produce mean increases in salivary cortisol. Psychoneuroendocrinology. 2009 Aug;34(7):953-67. doi: 10.1016/j.psyneuen.2009.02.010. Epub 2009 Mar 24. PMID 19321267

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT03830437/Prot_SAP_000.pdf